CLINICAL TRIAL: NCT02455609
Title: Intrathecally Administered Ketamine, Dexmedetomidine, and Their Combination With Bupivacaine for Postoperative Analgesia in Major Abdominal Cancer Surgery
Brief Title: Intrathecal Ketamine, Dexmedetomidine and Both With Bupivacaine for Postoperative Abdominal Cancer Surgery Pain
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd El-Rahman, Lecturer of anesthesia, intensive care, and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 210
Record Dates: First submitted 2015-05-18; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Therapy; Pain Management
Keywords: dexmedetomidine; ketamine; postoperative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Dexmedetomidine; Ketamine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- dexmedetomidine (I) (Active Comparator): intrathecal drug administartion of 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 5µg of dexmedetomidine in 1 ml volume.
  Interventions: Procedure: intrathecal drug administration; Drug: Dexmedetomidine; Drug: Bupivacaine
- ketamine (II) (Active Comparator): intrathecal drug administartion of 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 0.1 mg/kg ketamine in 1ml volume.
  Interventions: Procedure: intrathecal drug administration; Drug: ketamine; Drug: Bupivacaine
- Dexmedetomidine + Ketamine group (III) (Active Comparator): intrathecal drug administartion of patients in this arm received 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 5µg of dexmedetomidine plus 0.1 mg/kg of Ketamine in 1 ml volume.
  Interventions: Procedure: intrathecal drug administration; Drug: Dexmedetomidine; Drug: ketamine; Drug: Bupivacaine

INTERVENTIONS:
Procedure: intrathecal drug administration — pre-emptive intrathecal administration of analgesic medications for control of postoperative pain.
Drug: Dexmedetomidine
  Arms: Dexmedetomidine + Ketamine group (III); dexmedetomidine (I)
Drug: ketamine
  Arms: Dexmedetomidine + Ketamine group (III); ketamine (II)
Drug: Bupivacaine

SUMMARY:
Currently, opioids are widely used for pain relief, but they often provide sub-optimal analgesia with occasional serious side effects. Preservative-free ketamine hydrochloride was introduced as a spinal anesthetic more than twenty years ago and found to have advantages over local anesthetics. Intrathecal dexmedetomidine provides an analgesic effect in postoperative pain without severe sedation. The objectives of this study were to compare the efficacy and safety of intrathecally administered dexmedetomidine, ketamine, or their combination when added to bupivacaine for postoperative analgesia in major abdominal cancer surgery.

DETAILED DESCRIPTION:
This study was approved by the ethics committee of South Egypt Cancer Institute, Assiut University, Assiut, Egypt. After obtaining a written informed consent, 90 American Society of Anesthesia (ASA) I-II patients aged 30-50 years and scheduled for major abdominal cancer surgery were included in the study. Patients with a known allergy to the study drugs, significant cardiac, respiratory, renal or hepatic disease, coagulation disorder, infection at the site of intrathecal injection, drug or alcohol abuse, BMI > 30 kg/m2 , and psychiatric illnesses that would interfere with perception and assessment of pain were excluded from the study.

Preoperatively, patients were taught how to evaluate their own pain intensity using the visual analogue scale (VAS), scored from 0 -10 (where 0 = no pain, and 10 = the worst pain imaginable).

Oral diazepam (5 mg) was taken the night before surgery. Up on arrival at the operative theatre, a 16-gauge catheter was introduced intravenously at the dorsum of the hand; lactated Ringer's solution 10 mg/kg was infused intravenously over 10 min. before initiation of spinal anesthesia. Basic monitoring probes (electrocardiography, non invasive blood pressure, O2 saturation, and temperature) were applied. Patients were placed in the setting position and a 25-gauge Quincke needle was placed in the L2-3 or L3-4 interspaces.

Patients were randomly divided, by selecting sealed envelopes into one of three groups 30 patients each:

* The dexmedetomidine group (group I) received 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 5µg of dexmedetomidine in 1 ml volume intrathecally.
* The ketamine group (group II) received 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 0.1 mg/kg ketamine in 1ml volume intrathecally.
* Dexmedetomidine + Ketamine group (group III) received 10 mg of hyperbaric bupivacaine 0.5% in 2 ml volume and 5µg of dexmedetomidine plus 0.1 mg/kg of Ketamine in 1 ml volume intrathecally.

Immediately after their intrathecal injection, the patients were placed in the supine position. After successful spinal anesthesia, general anesthesia was induced with fentanyl 1.5-2 µg/kg, propofol 2-3 mg/kg, and lidocaine 1.5 mg/kg. Endotracheal intubation was facilitated by cis-atracurium 0.15 mg/kg. Heart rate, systolic, and diastolic blood pressure were recorded at 5, 10, 20, 30, 60, 120, 180 minutes. Anesthesia and muscle relaxation were maintained by isoflurane 1- 1.5 MAC in 50% oxygen/air mixture and cis-atracurium 0.03 mg/kg bolus given every 30 min. respectively.

At the end of surgery, muscle relaxation was reversed by neostigmine 50 µg/kg and atropine 20 µg/kg. Patients were extubated and transferred to postanesthesia care unit (PACU) and were monitored for vital signs (heart rate, non invasive blood pressure, respiratory rate, and O2 saturation) immediately postoperative and at 2, 4, 6, 12, 18, and 24 hours postoperative.

VAS scores were assessed at the same time points. Rescue analgesia represented by patient-controlled analgesia (PCA) with intravenous morphine with an initial bolus of 0.1 mg/kg once pain was expressed by the patient, or if VAS was 3 or more (VAS ≥ 3) followed by 1 mg boluses with a lockout period of 5 min. The time of first request of analgesia and total analgesic consumption in the first 24 hours postoperatively were recorded.

The patient's level of sedation was assessed at the same time points using a modified Observer's Assessment of alertness/sedation (OAAS) scale (where 6 = agitated, and 0 = doesn't respond to deep stimuls).

The attendant anesthesiologist, the patient-care giver, and the data collection personnel were all blinded to patient assignment to a specific group. Postoperative adverse effects such as nausea, vomiting, hypotension, bradycardia, cardiac arrhythmias were recorded and treated.

Hypotension was defined as a 15% decrease in systolic blood pressure from baseline. Bradycardia was defined as a heart rate slower than 50 beats per minute or a decrease in heart rate of 20% or more from baseline; whichever is lowest. Hypoxia was defined as an oxygen saturation of less than 90%. Hypotension was treated with intravenous boluse of ephidrine 0.1 mg/kg and normal saline 5ml/kg; the same doses were repeated as required. Bradycardia was treated with intravenous atropine 0.01 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-50 years
* American Society of Anesthesia (ASA) I-II patients
* scheduled for major abdominal cancer surgery

Exclusion Criteria:

* known allergy to the study drugs.
* significant cardiac, respiratory, renal or hepatic disease
* coagulation disorder
* infection at the site of intrathecal injection
* drug or alcohol abuse
* BMI > 30 kg/m2
* psychiatric illnesses that would interfere with perception and assessment of pain

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | the first 24 hours postoperative
  efficacy of analgesia

SECONDARY OUTCOMES:
time to first request of analgesia | the first 24 hours postoperative
  time needed by participating patients in each group to ask for rescue analgesia during the first 24 hours postoperative
total analgesic consumption | the first 24 hours postoperative
  total amount of rescue analgesic taken by patients in each group during the first 24 hours postoperative
side effects | the first 24 hours postoperative
  incidence of nausea (no.), vomiting (no.), hypotension (mmHg), bradycardia (b/m), hypertension (mmHg), arrhythmia (no.), sedation (by a 0-4 sedation scale) experienced by participating patients in each group

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Abd El-Rahman, M.D., Principal Investigator — South Egypt Cancer Institute, Assiut University, Egypt